CLINICAL TRIAL: NCT01533714
Title: Multi-center, Open-label, Follow-up Study to Assess the Long-term Safety and Efficacy of CDP6038 (Olokizumab) Administered Subcutaneously to Asian Subjects With Active Rheumatoid Arthritis Who Completed Study RA0083
Brief Title: The Long-term Safety and Efficacy of CDP6038 (Olokizumab) With Active Rheumatoid Arthritis
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Decision to out-license the compound for further development
Sponsor: UCB BIOSCIENCES, Inc. (Industry)
Collaborators: R-Pharm (Industry)
Responsible Party: Sponsor
Organization: UCB Pharma (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RA0089
Record Dates: First submitted 2012-02-10; First posted 2012-02-15 (Estimated); Results first posted 2022-05-17 (Actual); Last update posted 2022-05-20 (Actual); Status verified 2022-05

CONDITIONS: Rheumatoid Arthritis
Keywords: Rheumatoid Arthritis; Monoclonal antibody; Interleukin-6; Olokizumab; CDP6038
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — olokizumab

STUDY DESIGN:
Intervention Model Description: RA0089 is a single arm study, however, analysis will also be performed according to the original treatment arms of the parent study NCT01463059 (RA0083).
Oversight: Data Monitoring Committee: No

ARMS (1):
- CDP6038 (olokizumab) (Experimental): CDP6038 (olokizumab) 120 mg: subcutaneous injections at q2w (every two weeks). RA0089 is a single arm study, however, analysis will be presented according to the original treatment arms of the parent study NCT01463059 (RA0083).
  Interventions: Biological: CDP6038 (olokizumab)

INTERVENTIONS:
Biological: CDP6038 (olokizumab) — Biological/Vaccine: CDP6038 (olokizumab) 100 mg/mL solution for subcutaneous (sc) injection

SUMMARY:
The purpose of this study is to evaluate the long-term safety and tolerability of CDP6038 (olokizumab) treatment in adult subjects with active rheumatoid arthritis (RA) who completed study RA0083 [NCT01463059].

DETAILED DESCRIPTION:
Male and female subjects were randomized in a multi-center, open-label, follow-up study to assess the long-term safety and efficacy of a subcutaneous dose of 120 mg CDP6038 (olokizumab), every 2 weeks (q2w), for the treatment of active RA.

ELIGIBILITY:
Inclusion Criteria:

* Completed the RA0083 [NCT01463059] study (Week 12 Visit)
* Must have maintained their stable dose (and route) of methotrexate (MTX) between 6 to 16 mg/week in Japan or 7.5 to 20 mg/week in Korea and Taiwan in RA0083 [NCT01463059], and plan to maintain this same dose and route of administration for at least 12 weeks
* Female subjects must be either postmenopausal for at least 1 year, surgically incapable of childbearing, or effectively practicing 2 acceptable methods of contraception

Exclusion Criteria:

* Have an ongoing SAE from the RA0083 [NCT01463059] study
* Female subjects who are breast-feeding, pregnant, or plan to become pregnant during the study or within 24 weeks
* Have evidence of active or latent tuberculosis (TB)
* Subject is receiving any biologic response modifier or synthetic disease-modifying antirheumatic drug (DMARD) other than MTX
* Subject has planned surgery during the first 12 weeks of the study
* Subjects who tested positive for hepatitis B core antibody (HBcAb) and/or hepatitis B surface antibody (HBsAb) at Screening in RA0083 [NCT01463059] and who subsequently test positive for hepatitis B virus deoxyribonucleic acid (HBV DNA) at Week 12 of RA0083 [NCT01463059]

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 103 (Actual)
Dates: Start 2012-01-26 (Actual); Primary Completion 2013-11-27 (Actual); Study Completion 2013-11-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tsutomu Takeuchi, Professor, Principal Investigator — Keio University
Locations (32):
- Japan (21):
  - 102, Chiba
  - 114, Fukuoka
  - 115, Fukuoka
  - 113, Hiroshima
  - 120, Kakogawa
  - 118, Kumamoto
  - 116, Kurume
  - 122, Matsuyama
  - 107, Nagaoka
  - 110, Nagoya
  - 103, Narita
  - 112, Okayama
  - 119, Ōita
  - 100, Sapporo
  - 117, Sasebo
  - 123, Tokyo
  - 101, Tomakomai
  - 108, Tonami
  - 111, Tsu
  - 105, Yokohama
  - 104, Yotukaido
- South Korea (5):
  - 200, Daejeon
  - 201, Junggu
  - 202, Seongdong-Gu
  - 203, Seoul
  - 204, Seoul
- Taiwan (6):
  - 301, Taichung
  - 306, Taichung
  - 307, Taichung
  - 302, Taipei
  - 308, Taipei
  - 309, Taipei

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The present study was an open-label extension to study RA0083 (NCT01463059). Subjects completing the 12-week treatment period of study RA0083 had the opportunity to participate in this study. First subject enrolled: 26 January 2012. Last subject completed: 27 November 2013.
Pre-assignment Details: 105 subjects completed the parent Study RA0083 (NCT01463059); 103 subjects were enrolled in Study RA0089.
Groups:
- RA0083 CDP6038 (Olokizumab) 120 mg q2w: CDP6038 (olokizumab) 120 mg administered q2w sc in Study RA0083, and maintained at same dose (i.e. 120 mg q2w sc) at start of Study RA0089 (Week 12 of RA0083).
- RA0083 CDP6038 (Olokizumab) 120 mg q4w: CDP6038 (olokizumab) 120 mg administered every 4 weeks (q4w) sc in Study RA0083, followed by switch to CDP6038 (olokizumab) 120 mg q2w sc at start of Study RA0089 (Week 12 of RA0083).
- RA0083 CDP6038 (Olokizumab) 240 mg q4w: CDP6038 (olokizumab) 240 mg administered q4w sc in Study RA0083, followed by switch to CDP6038 (olokizumab) 120 mg q2w sc at start of Study RA0089 (Week 12 of RA0083).
- RA0083 CDP6038 (Olokizumab) 60 mg q2w: CDP6038 (olokizumab) 60 mg administered q2w sc in Study RA0083, followed by switch to CDP6038 (olokizumab) 120 mg q2w sc at start of Study RA0089 (Week 12 of RA0083).
- RA0083 CDP6038 (Olokizumab) 60 mg q4w: CDP6038 (olokizumab) 60 mg administered q4w sc in Study RA0083, followed by switch to CDP6038 (olokizumab) 120 mg q2w sc at start of Study RA0089 (Week 12 of RA0083).
- RA0083 Placebo: Placebo (sodium chloride, 0.9%) was administered sc in Study RA0083, followed by switch to CDP6038 (olokizumab) 120 mg q2w sc at start of Study RA0089 (Week 12 of RA0083).
Period: Overall Study
Arm/Group | RA0083 CDP6038 (Olokizumab) 120 mg q2w | RA0083 CDP6038 (Olokizumab) 120 mg q4w | RA0083 CDP6038 (Olokizumab) 240 mg q4w | RA0083 CDP6038 (Olokizumab) 60 mg q2w | RA0083 CDP6038 (Olokizumab) 60 mg q4w | RA0083 Placebo
Started | 10 | 15 | 11 | 15 | 28 | 24
Completed | 10 | 12 | 7 | 11 | 21 | 21
Not Completed | 0 | 3 | 4 | 4 | 7 | 3
Not completed — Adverse Event | 0 | 1 | 2 | 2 | 2 | 1
Not completed — Lack of Efficacy | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1 | 0 | 1 | 1 | 0
Not completed — Exclusion criteria | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Positive for purified protein derivative | 0 | 0 | 1 | 0 | 1 | 0
Not completed — Withdrawal criteria | 0 | 0 | 1 | 0 | 3 | 1
Not completed — Ineligibility reason | 0 | 0 | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Safety Population included all enrolled subjects who received at least 1 injection of CDP6038 (olokizumab) in Study RA0089.
Groups:
- RA0083 CDP6038 (Olokizumab) 120 mg q4w: CDP6038 (olokizumab) 120 mg administered q4w sc in Study RA0083, followed by switch to CDP6038 (olokizumab) 120 mg q2w sc at start of Study RA0089 (Week 12 of RA0083).
- Total: Total of all reporting groups
Arm/Group | RA0083 CDP6038 (Olokizumab) 120 mg q2w | RA0083 CDP6038 (Olokizumab) 120 mg q4w | RA0083 CDP6038 (Olokizumab) 240 mg q4w | RA0083 CDP6038 (Olokizumab) 60 mg q2w | RA0083 CDP6038 (Olokizumab) 60 mg q4w | RA0083 Placebo | Total
Number analyzed (Participants) | 10 | 15 | 11 | 15 | 28 | 24 | 103
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 7 | 11 | 10 | 13 | 23 | 18 | 82
  >=65 years | 3 | 4 | 1 | 2 | 5 | 6 | 21
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 12 | 9 | 12 | 27 | 21 | 88
  Male | 3 | 3 | 2 | 3 | 1 | 3 | 15

OUTCOME MEASURES:

1. Primary Outcome: Total Number of Subjects With Treatment-emergent Adverse Events (TEAEs)
Description: Reported TEAEs included adverse events that started or worsened after the first dose of CDP6038 (olokizumab) in Study RA0089 and within 30 days after the last dose.
Time Frame: From Baseline (Week 0 of Study RA0089) until 30 days after the last dose (maximum up to 562 days)
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | RA0083 CDP6038 (Olokizumab) 120 mg q2w | RA0083 CDP6038 (Olokizumab) 120 mg q4w | RA0083 CDP6038 (Olokizumab) 240 mg q4w | RA0083 CDP6038 (Olokizumab) 60 mg q2w | RA0083 CDP6038 (Olokizumab) 60 mg q4w | RA0083 Placebo
Number analyzed (Participants) | 10 | 15 | 11 | 15 | 28 | 24
Participants | 8 | 13 | 10 | 12 | 25 | 22

2. Secondary Outcome: Change From Baseline (Week 0 of Study RA0083) in the Disease Activity Score-28-joint Count (C-reactive Protein) (DAS28[CRP]) at Week 12 of Study RA0089
Description: DAS28(CRP) was calculated using tender/painful joint count (TJC) and swollen joint count (SJC) from 28 joints, Patient's Global Assessment of Disease Activity (PtGADA)-Visual Analog Scale (VAS), and CRP as per formula: DAS28(CRP)=0.56 * (TJC)^1/2 + 0.28 * (SJC)^1/2 + 0.36 * ln(CRP[mg/L]+1) + 0.014 * PtGADA + 0.96 Assessments: •TJC and SJC: assessed on same 2-point scale (0=absent; 1=present). • PtGADA: 100 mm VAS (0=very good, no symptoms; 100=very poor, severe symptoms). • CRP value calculated in mg/L. 28 joints included shoulders, elbows, wrists; metacarpophalangeal (MCP), thumb interphalangeal (IP), and proximal interphalangeal (PIP) joints of hands; and knees. Scores on DAS28(CRP) range from 0 to approximately 10, where scores greater than (>) 5.1 correspond with active disease, scores less than (<) 3.2 correspond with well controlled disease, and scores <2.6 correspond with remission or similar. A negative change in DAS28(CRP) score indicates an improvement in disease activity.
Time Frame: Baseline (Week 0 of Study RA0083) and Week 12 (Study RA0089)
Population: Full Analysis Set (FAS) included all enrolled subjects who received at least 1 injection of CDP6038 (olokizumab) and in addition had at least 1 efficacy measurement in Study RA0089. Here, number of participants analyzed included all participants who were evaluable for this outcome measure (assessed at Baseline and postbaseline timepoint).
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | RA0083 CDP6038 (Olokizumab) 120 mg q2w | RA0083 CDP6038 (Olokizumab) 120 mg q4w | RA0083 CDP6038 (Olokizumab) 240 mg q4w | RA0083 CDP6038 (Olokizumab) 60 mg q2w | RA0083 CDP6038 (Olokizumab) 60 mg q4w | RA0083 Placebo
Number analyzed (Participants) | 10 | 14 | 10 | 13 | 23 | 23
units on a scale | -2.9618 (1.05692) | -2.5358 (1.11550) | -2.9758 (1.23346) | -2.7948 (1.28792) | -2.6837 (0.80614) | -2.5902 (1.06296)

3. Secondary Outcome: Change From Baseline (Week 0 of Study RA0083) in DAS28(CRP) at Week 24 of Study RA0089
Description: DAS28(CRP) was calculated using the TJC and SJC from 28 joints, the PtGADA-VAS, andCRP according to the formula: DAS28(CRP)=0.56 * (TJC)^1/2 + 0.28 * (SJC)^1/2 + 0.36 * ln(CRP[mg/L]+1) + 0.014 * PtGADA + 0.96 Assessments: • TJC and SJC: assessed on same 2-point scale (0=absent; 1=present). • PtGADA: 100 mm VAS (0=very good, no symptoms; 100=very poor, severe symptoms). • CRP value calculated in mg/L. The 28 joints included shoulders, elbows, wrists; MCP, thumb IP, and PIP joints of hands; and knees. Scores on DAS28(CRP) range from 0 to approximately 10, where scores >5.1 correspond with active disease, scores <3.2 correspond with well controlled disease, and scores <2.6 correspond with remission or similar. A negative change in DAS28(CRP) score indicates an improvement in disease activity.
Time Frame: Baseline (Week 0 of Study RA0083) and Week 24 (Study RA0089)
Population: FAS included all enrolled subjects who received at least 1 injection of CDP6038 (olokizumab) and in addition had at least 1 efficacy measurement in Study RA0089. Here, number of participants analyzed included all participants who were evaluable for this outcome measure (assessed at Baseline and postbaseline timepoint).
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | RA0083 CDP6038 (Olokizumab) 120 mg q2w | RA0083 CDP6038 (Olokizumab) 120 mg q4w | RA0083 CDP6038 (Olokizumab) 240 mg q4w | RA0083 CDP6038 (Olokizumab) 60 mg q2w | RA0083 CDP6038 (Olokizumab) 60 mg q4w | RA0083 Placebo
Number analyzed (Participants) | 8 | 9 | 10 | 11 | 22 | 22
units on a scale | -2.6916 (0.75807) | -3.3277 (1.05841) | -3.3523 (0.74516) | -2.8884 (1.43276) | -3.0176 (0.82217) | -2.8235 (0.99271)

4. Secondary Outcome: Change From Baseline (Week 0 of Study RA0083) in DAS28(CRP) at Week 48 of Study RA0089
Description: as for outcome 3
Time Frame: Baseline (Week 0 of Study RA0083) and Week 48 (Study RA0089)
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | RA0083 CDP6038 (Olokizumab) 120 mg q2w | RA0083 CDP6038 (Olokizumab) 120 mg q4w | RA0083 CDP6038 (Olokizumab) 240 mg q4w | RA0083 CDP6038 (Olokizumab) 60 mg q2w | RA0083 CDP6038 (Olokizumab) 60 mg q4w | RA0083 Placebo
Number analyzed (Participants) | 3 | 3 | 6 | 4 | 7 | 9
units on a scale | -2.6243 (1.52735) | -3.2720 (0.97343) | -3.2397 (0.85356) | -2.9625 (1.16236) | -2.4750 (1.31771) | -3.2211 (0.45471)

5. Secondary Outcome: Change From Baseline (Week 0 of Study RA0083) in DAS28(CRP) at Week 96 of Study RA0089
Description: DAS28(CRP) was calculated using the TJC and SJC from 28 joints, the PtGADA-VAS, andCRP according to the formula: DAS28(CRP)=0.56 * (TJC)^1/2 + 0.28 * (SJC)^1/2 + 0.36 * ln(CRP[mg/L]+1) + 0.014 * PtGADA + 0.96 Assessments: • TJC and SJC: assessed on same 2-point scale (0=absent; 1=present). • PtGADA: 100 mm VAS (0=very good, no symptoms; 100=very poor, severe symptoms). • CRP value calculated in mg/L. The 28 joints included shoulders, elbows, wrists; MCP, thumb IP, and PIP joints of hands; and knees. Scores on DAS28(CRP) range from 0 to approximately 10, where scores >5.1 correspond with active disease, scores <3.2 correspond with well controlled disease, and scores <2.6 correspond with remission or similar. A negative change in DAS28(CRP) score indicates an improvement in disease activity. Since the study was terminated early before Week 96, no results data are available for analysis at the Week 96 time point and this Outcome Measure has zero total participants analyzed.
Time Frame: Baseline (Week 0 of Study RA0083) and Week 96 (Study RA0089)
Reporting Status: Not Posted

6. Secondary Outcome: The American College of Rheumatology (ACR) 20% (ACR20) Improvement Criteria Response Rate From Baseline (Week 0 of Study RA0083) at Week 12 of Study RA0089
Description: ACR20 represents at least 20% improvement from Baseline in TJC (68 joints) + in SJC (66 joints) + in at least 3 of 5 core set measures: PtGADA-VAS, Physician's Global Assessment of Disease Activity (PhGADA)-VAS, Patient's Assessment of Arthritis Pain (PAAP)-VAS, Health Assessment Questionnaire-Disability Index (HAQ-DI) and CRP. Assessments: • TJC and SJC: same 2-point scale (0=absent;1=present). • PtGADA: 100 mm VAS (0=very good, no symptoms;100=very poor, severe symptoms). • PhGADA: 100 mm VAS (0=very good, asymptomatic, no limitation of normal activities;100=very poor, very severe symptoms which were intolerable, inability to carry out all normal activities). • PAAP: 100 mm VAS (0=no pain;100=most severe pain). • HAQ-DI assessed degree of difficulty experienced in 8 domains of daily living activities (20 questions), total score (0-3) computed from item scores, with lower scores meaning less disability. • CRP in mg/L. Missing values were considered as non-responding status.
Time Frame: Baseline (Week 0 of Study RA0083) and Week 12 (Study RA0089)
Population: FAS included all enrolled subjects who received at least 1 injection of CDP6038 (olokizumab) and in addition had at least 1 efficacy measurement in Study RA0089.
Measure: Number; unit: Percentage of responders
Arm/Group | RA0083 CDP6038 (Olokizumab) 120 mg q2w | RA0083 CDP6038 (Olokizumab) 120 mg q4w | RA0083 CDP6038 (Olokizumab) 240 mg q4w | RA0083 CDP6038 (Olokizumab) 60 mg q2w | RA0083 CDP6038 (Olokizumab) 60 mg q4w | RA0083 Placebo
Number analyzed (Participants) | 10 | 15 | 11 | 14 | 28 | 24
Percentage of responders | 100.0 | 60.0 | 81.8 | 71.4 | 64.3 | 70.8

7. Secondary Outcome: The ACR20 Improvement Criteria Response Rate From Baseline (Week 0 of Study RA0083) at Week 24 of Study RA0089
Description: ACR20 represents at least 20% improvement from Baseline in TJC (68 joints) + SJC (66 joints) + in at least 3 of 5 core set measures: PtGADA-VAS, PhGADA-VAS, PAAP-VAS, HAQ-DI and CRP. Assessments: • TJC and SJC: same 2-point scale (0=absent;1=present). • PtGADA: 100 mm VAS (0=very good, no symptoms;100=very poor, severe symptoms). • PhGADA: 100 mm VAS (0=very good, asymptomatic, no limitation of normal activities;100=very poor, very severe symptoms which were intolerable, inability to carry out all normal activities). • PAAP: 100 mm VAS (0=no pain;100=most severe pain). • HAQ-DI assessed degree of difficulty experienced in 8 domains of daily living activities (20 questions), total score (0-3) computed from item scores, with lower scores meaning less disability. • CRP in mg/L. Missing values were considered as non-responding status.
Time Frame: Baseline (Week 0 of Study RA0083) and Week 24 (Study RA0089)
Population: as for outcome 6
Measure: Number; unit: Percentage of responders
Arm/Group | RA0083 CDP6038 (Olokizumab) 120 mg q2w | RA0083 CDP6038 (Olokizumab) 120 mg q4w | RA0083 CDP6038 (Olokizumab) 240 mg q4w | RA0083 CDP6038 (Olokizumab) 60 mg q2w | RA0083 CDP6038 (Olokizumab) 60 mg q4w | RA0083 Placebo
Number analyzed (Participants) | 10 | 15 | 11 | 14 | 28 | 24
Percentage of responders | 60.0 | 46.7 | 81.8 | 57.1 | 71.4 | 66.7

8. Secondary Outcome: The ACR20 Improvement Criteria Response Rate From Baseline (Week 0 of Study RA0083) at Week 48 of Study RA0089
Description: as for outcome 7
Time Frame: Baseline (Week 0 of Study RA0083) and Week 48 (Study RA0089)
Population: as for outcome 6
Measure: Number; unit: Percentage of responders
Arm/Group | RA0083 CDP6038 (Olokizumab) 120 mg q2w | RA0083 CDP6038 (Olokizumab) 120 mg q4w | RA0083 CDP6038 (Olokizumab) 240 mg q4w | RA0083 CDP6038 (Olokizumab) 60 mg q2w | RA0083 CDP6038 (Olokizumab) 60 mg q4w | RA0083 Placebo
Number analyzed (Participants) | 10 | 15 | 11 | 14 | 28 | 24
Percentage of responders | 20.0 | 13.3 | 54.5 | 21.4 | 21.4 | 33.3

9. Secondary Outcome: The ACR20 Improvement Criteria Response Rate From Baseline (Week 0 of Study RA0083) at Week 96 of Study RA0089
Description: ACR20: at least 20% improvement from Baseline in TJC (68 joints) + SJC (66 joints) + in at least 3 of 5 core set measures: PtGADA-VAS, PhGADA-VAS, PAAP-VAS, HAQ-DI and CRP. Assessments: • TJC and SJC: same 2-point scale (0=absent;1=present). • PtGADA: 100 mm VAS (0=very good, no symptoms;100=very poor, severe symptoms). • PhGADA: 100 mm VAS (0=very good, asymptomatic, no limitation of normal activities;100=very poor, very severe symptoms which were intolerable, inability to carry out all normal activities). • PAAP: 100 mm VAS (0=no pain;100=most severe pain). • HAQ-DI assessed degree of difficulty experienced in 8 domains of daily living activities (20 questions), total score (0-3) computed from item scores, with lower scores meaning less disability. • CRP in mg/L. Missing values were considered as non-responding status. Since the study was terminated early before Week 96, no data was collected and analyzed at the Week 96 and this Outcome Measure has zero total participants analyzed.
Time Frame: Baseline (Week 0 of Study RA0083) and Week 96 (Study RA0089)
Reporting Status: Not Posted

10. Secondary Outcome: The ACR 50% (ACR50) Improvement Criteria Response Rate From Baseline (Week 0 of Study RA0083) at Week 12 of Study RA0089
Description: ACR50 represents at least 50% improvement from Baseline in TJC (68 joints) + in SJC (66 joints) + in at least 3 of 5 core set measures: PtGADA-VAS, PhGADA-VAS, PAAP-VAS, HAQ-DI and CRP. Assessments: • TJC and SJC: same 2-point scale (0=absent;1=present). • PtGADA: 100 mm VAS (0=very good, no symptoms;100=very poor, severe symptoms). • PhGADA: 100 mm VAS (0=very good, asymptomatic, no limitation of normal activities;100=very poor, very severe symptoms which were intolerable, inability to carry out all normal activities). • PAAP: 100 mm VAS (0=no pain;100=most severe pain). • HAQ-DI assessed degree of difficulty experienced in 8 domains of daily living activities (20 questions), total score (0-3) computed from item scores, with lower scores meaning less disability. • CRP in mg/L. Missing values were considered as non-responding status.
Time Frame: Baseline (Week 0 of Study RA0083) and Week 12 (Study RA0089)
Population: as for outcome 6
Measure: Number; unit: Percentage of responders
Arm/Group | RA0083 CDP6038 (Olokizumab) 120 mg q2w | RA0083 CDP6038 (Olokizumab) 120 mg q4w | RA0083 CDP6038 (Olokizumab) 240 mg q4w | RA0083 CDP6038 (Olokizumab) 60 mg q2w | RA0083 CDP6038 (Olokizumab) 60 mg q4w | RA0083 Placebo
Number analyzed (Participants) | 10 | 15 | 11 | 14 | 28 | 24
Percentage of responders | 70.0 | 40.0 | 54.5 | 42.9 | 42.9 | 50.0

11. Secondary Outcome: The ACR50 Improvement Criteria Response Rate From Baseline (Week 0 of Study RA0083) at Week 24 of Study RA0089
Description: as for outcome 10
Time Frame: Baseline (Week 0 of Study RA0083) and Week 24 (Study RA0089)
Population: as for outcome 6
Measure: Number; unit: Percentage of responders
Arm/Group | RA0083 CDP6038 (Olokizumab) 120 mg q2w | RA0083 CDP6038 (Olokizumab) 120 mg q4w | RA0083 CDP6038 (Olokizumab) 240 mg q4w | RA0083 CDP6038 (Olokizumab) 60 mg q2w | RA0083 CDP6038 (Olokizumab) 60 mg q4w | RA0083 Placebo
Number analyzed (Participants) | 10 | 15 | 11 | 14 | 28 | 24
Percentage of responders | 40.0 | 40.0 | 63.6 | 57.1 | 42.9 | 45.8

12. Secondary Outcome: The ACR50 Improvement Criteria Response Rate From Baseline (Week 0 of Study RA0083) at Week 48 of Study RA0089
Description: as for outcome 10
Time Frame: Baseline (Week 0 of Study RA0083) and Week 48 (Study RA0089)
Population: as for outcome 6
Measure: Number; unit: Percentage of responders
Arm/Group | RA0083 CDP6038 (Olokizumab) 120 mg q2w | RA0083 CDP6038 (Olokizumab) 120 mg q4w | RA0083 CDP6038 (Olokizumab) 240 mg q4w | RA0083 CDP6038 (Olokizumab) 60 mg q2w | RA0083 CDP6038 (Olokizumab) 60 mg q4w | RA0083 Placebo
Number analyzed (Participants) | 10 | 15 | 11 | 14 | 28 | 24
Percentage of responders | 20.0 | 13.3 | 45.5 | 14.3 | 17.9 | 29.2

13. Secondary Outcome: The ACR50 Improvement Criteria Response Rate From Baseline (Week 0 of Study RA0083) at Week 96 of Study RA0089
Description: ACR50:atleast 50% improvement from Baseline in TJC (68 joints) + in SJC (66 joints) + in at least 3 of 5 core set measures: PtGADA-VAS, PhGADA-VAS, PAAP-VAS, HAQ-DI and CRP. Assessments: • TJC and SJC: same 2-point scale (0=absent;1=present). • PtGADA: 100 mm VAS (0=very good, no symptoms;100=very poor, severe symptoms). • PhGADA: 100 mm VAS (0=very good, asymptomatic, no limitation of normal activities;100=very poor, very severe symptoms which were intolerable, inability to carry out all normal activities). • PAAP: 100 mm VAS (0=no pain;100=most severe pain). • HAQ-DI assessed degree of difficulty experienced in 8 domains of daily living activities (20 questions), total score (0-3) computed from item scores, with lower scores meaning less disability. • CRP in mg/L. Missing values were considered as non-responding status. Since the study was terminated early before Week 96, no data was collected and analyzed at the Week 96 and this Outcome Measure has zero total participants analyzed.
Time Frame: Baseline (Week 0 of Study RA0083) and Week 96 (Study RA0089)
Reporting Status: Not Posted

14. Secondary Outcome: The ACR 70% (ACR70) Improvement Criteria Response Rate From Baseline (Week 0 of Study RA0083) at Week 12 of Study RA0089
Description: ACR70 represents at least 70% improvement from Baseline in TJC (68 joints) + in SJC (66 joints) + in at least 3 of 5 core set measures: PtGADA-VAS, PhGADA-VAS, PAAP-VAS, HAQ-DI and CRP. Assessments: • TJC and SJC: same 2-point scale (0=absent;1=present). • PtGADA: 100 mm VAS (0=very good, no symptoms;100=very poor, severe symptoms). • PhGADA: 100 mm VAS (0=very good, asymptomatic, no limitation of normal activities;100=very poor, very severe symptoms which were intolerable, inability to carry out all normal activities). • PAAP: 100 mm VAS (0=no pain;100=most severe pain). • HAQ-DI assessed degree of difficulty experienced in 8 domains of daily living activities (20 questions), total score (0-3) computed from item scores, with lower scores meaning less disability. • CRP in mg/L. Missing values were considered as non-responding status.
Time Frame: Baseline (Week 0 of Study RA0083) and Week 12 (Study RA0089)
Population: as for outcome 6
Measure: Number; unit: Percentage of responders
Arm/Group | RA0083 CDP6038 (Olokizumab) 120 mg q2w | RA0083 CDP6038 (Olokizumab) 120 mg q4w | RA0083 CDP6038 (Olokizumab) 240 mg q4w | RA0083 CDP6038 (Olokizumab) 60 mg q2w | RA0083 CDP6038 (Olokizumab) 60 mg q4w | RA0083 Placebo
Number analyzed (Participants) | 10 | 15 | 11 | 14 | 28 | 24
Percentage of responders | 30.0 | 26.7 | 27.3 | 21.4 | 17.9 | 29.2

15. Secondary Outcome: The ACR70 Improvement Criteria Response Rate From Baseline (Week 0 of Study RA0083) at Week 24 of Study RA0089
Description: as for outcome 14
Time Frame: Baseline (Week 0 of Study RA0083) and Week 24 (Study RA0089)
Population: as for outcome 6
Measure: Number; unit: Percentage of responders
Arm/Group | RA0083 CDP6038 (Olokizumab) 120 mg q2w | RA0083 CDP6038 (Olokizumab) 120 mg q4w | RA0083 CDP6038 (Olokizumab) 240 mg q4w | RA0083 CDP6038 (Olokizumab) 60 mg q2w | RA0083 CDP6038 (Olokizumab) 60 mg q4w | RA0083 Placebo
Number analyzed (Participants) | 10 | 15 | 11 | 14 | 28 | 24
Percentage of responders | 10.0 | 20.0 | 54.5 | 42.9 | 32.1 | 25.0

16. Secondary Outcome: The ACR70 Improvement Criteria Response Rate From Baseline (Week 0 of Study RA0083) at Week 48 of Study RA0089
Description: as for outcome 14
Time Frame: Baseline (Week 0 of Study RA0083) and Week 48 (Study RA0089)
Population: as for outcome 6
Measure: Number; unit: Percentage of responders
Arm/Group | RA0083 CDP6038 (Olokizumab) 120 mg q2w | RA0083 CDP6038 (Olokizumab) 120 mg q4w | RA0083 CDP6038 (Olokizumab) 240 mg q4w | RA0083 CDP6038 (Olokizumab) 60 mg q2w | RA0083 CDP6038 (Olokizumab) 60 mg q4w | RA0083 Placebo
Number analyzed (Participants) | 10 | 15 | 11 | 14 | 28 | 24
Percentage of responders | 10.0 | 13.3 | 18.2 | 14.3 | 7.1 | 16.7

17. Secondary Outcome: The ACR70 Improvement Criteria Response Rate From Baseline (Week 0 of Study RA0083) at Week 96 of Study RA0089
Description: ACR70:atleast 70% improvement from Baseline in TJC (68 joints) + in SJC (66 joints) + in at least 3 of 5 core set measures: PtGADA-VAS, PhGADA-VAS, PAAP-VAS, HAQ-DI and CRP. Assessments: • TJC and SJC: same 2-point scale (0=absent;1=present). • PtGADA: 100 mm VAS (0=very good, no symptoms;100=very poor, severe symptoms). • PhGADA: 100 mm VAS (0=very good, asymptomatic, no limitation of normal activities;100=very poor, very severe symptoms which were intolerable, inability to carry out all normal activities). • PAAP: 100 mm VAS (0=no pain;100=most severe pain). • HAQ-DI assessed degree of difficulty experienced in 8 domains of daily living activities (20 questions), total score (0-3) computed from item scores, with lower scores meaning less disability. • CRP in mg/L. Missing values were considered as non-responding status. Since the study was terminated early before Week 96, no data was collected and analyzed at the Week 96 and this Outcome Measure has zero total participants analyzed.
Time Frame: Baseline (Week 0 of Study RA0083) and Week 96 (Study RA0089)
Reporting Status: Not Posted

18. Secondary Outcome: Percentage of Subjects With DAS28(CRP) <2.6 at Week 12 of Study RA0089
Description: DAS28(CRP) was calculated using the TJC and SJC from 28 joints, the PtGADA-VAS, andCRP according to the formula: DAS28(CRP)=0.56 * (TJC)^1/2 + 0.28 * (SJC)^1/2 + 0.36 * ln(CRP[mg/L]+1) + 0.014 * PtGADA + 0.96 Assessments: • TJC and SJC: assessed on same 2-point scale (0=absent; 1=present). • PtGADA: 100 mm VAS (0=very good, no symptoms; 100=very poor, severe symptoms). • CRP value calculated in mg/L. The 28 joints included shoulders, elbows, wrists; MCP, thumb IP, and PIP joints of hands; and knees. Scores on DAS28(CRP) range from 0 to approximately 10, where scores >5.1 correspond with active disease, scores <3.2 correspond with well controlled disease, and scores <2.6 correspond with remission or similar. Percentage of participants with DAS28(CRP) <2.6 were reported.
Time Frame: Week 12 (Study RA0089)
Population: as for outcome 6
Measure: Number; unit: Percentage of subjects
Arm/Group | RA0083 CDP6038 (Olokizumab) 120 mg q2w | RA0083 CDP6038 (Olokizumab) 120 mg q4w | RA0083 CDP6038 (Olokizumab) 240 mg q4w | RA0083 CDP6038 (Olokizumab) 60 mg q2w | RA0083 CDP6038 (Olokizumab) 60 mg q4w | RA0083 Placebo
Number analyzed (Participants) | 10 | 15 | 11 | 14 | 28 | 24
Percentage of subjects | 50.00 | 64.29 | 70.00 | 53.85 | 43.48 | 39.13

19. Secondary Outcome: Percentage of Subjects With DAS28(CRP) <2.6 at Week 24 of Study RA0089
Description: as for outcome 18
Time Frame: Week 24 (Study RA0089)
Population: as for outcome 6
Measure: Number; unit: Percentage of subjects
Arm/Group | RA0083 CDP6038 (Olokizumab) 120 mg q2w | RA0083 CDP6038 (Olokizumab) 120 mg q4w | RA0083 CDP6038 (Olokizumab) 240 mg q4w | RA0083 CDP6038 (Olokizumab) 60 mg q2w | RA0083 CDP6038 (Olokizumab) 60 mg q4w | RA0083 Placebo
Number analyzed (Participants) | 10 | 15 | 11 | 14 | 28 | 24
Percentage of subjects | 50.00 | 77.78 | 80.00 | 54.55 | 59.09 | 40.91

20. Secondary Outcome: Percentage of Subjects With DAS28(CRP) <2.6 at Week 48 of Study RA0089
Description: as for outcome 18
Time Frame: Week 48 (Study RA0089)
Population: as for outcome 6
Measure: Number; unit: Percentage of subjects
Arm/Group | RA0083 CDP6038 (Olokizumab) 120 mg q2w | RA0083 CDP6038 (Olokizumab) 120 mg q4w | RA0083 CDP6038 (Olokizumab) 240 mg q4w | RA0083 CDP6038 (Olokizumab) 60 mg q2w | RA0083 CDP6038 (Olokizumab) 60 mg q4w | RA0083 Placebo
Number analyzed (Participants) | 10 | 15 | 11 | 14 | 28 | 24
Percentage of subjects | 66.67 | 100.00 | 83.33 | 100.00 | 42.86 | 55.56

21. Secondary Outcome: Percentage of Subjects With DAS28(CRP) <2.6 at Week 96 of Study RA0089
Description: DAS28(CRP) was calculated using the TJC and SJC from 28 joints, the PtGADA-VAS, andCRP according to the formula: DAS28(CRP)=0.56 * (TJC)^1/2 + 0.28 * (SJC)^1/2 + 0.36 * ln(CRP[mg/L]+1) + 0.014 * PtGADA + 0.96 Assessments: • TJC and SJC: assessed on same 2-point scale (0=absent; 1=present). • PtGADA: 100 mm VAS (0=very good, no symptoms; 100=very poor, severe symptoms). • CRP value calculated in mg/L. The 28 joints included shoulders, elbows, wrists; MCP, thumb IP, and PIP joints of hands; and knees. Scores on DAS28(CRP) range from 0 to approximately 10, where scores >5.1 correspond with active disease, scores <3.2 correspond with well controlled disease, and scores <2.6 correspond with remission or similar. Percentage of participants with DAS28(CRP) <2.6 were reported. Since the study was terminated early before Week 96, no data was collected and analyzed at the Week 96 and this Outcome Measure has zero total participants analyzed.
Time Frame: Week 96 (Study RA0089)
Reporting Status: Not Posted

22. Secondary Outcome: Percentage of Subjects With DAS28(CRP) ≤3.2 at Week 12 of Study RA0089
Description: DAS28(CRP) was calculated using the TJC and SJC from 28 joints, the PtGADA-VAS, andCRP according to the formula: DAS28(CRP)=0.56 * (TJC)^1/2 + 0.28 * (SJC)^1/2 + 0.36 * ln(CRP[mg/L]+1) + 0.014 * PtGADA + 0.96 Assessments: • TJC and SJC: assessed on same 2-point scale (0=absent; 1=present). • PtGADA: 100 mm VAS (0=very good, no symptoms; 100=very poor, severe symptoms). • CRP value calculated in mg/L. The 28 joints included shoulders, elbows, wrists; MCP, thumb IP, and PIP joints of hands; and knees. Scores on DAS28(CRP) range from 0 to approximately 10, where scores >5.1 correspond with active disease, scores <3.2 correspond with well controlled disease, and scores <2.6 correspond with remission or similar. Percentage of participants with DAS28(CRP) less than or equal to (≤) 3.2 were reported.
Time Frame: Week 12 (Study RA0089)
Population: as for outcome 6
Measure: Number; unit: Percentage of subjects
Arm/Group | RA0083 CDP6038 (Olokizumab) 120 mg q2w | RA0083 CDP6038 (Olokizumab) 120 mg q4w | RA0083 CDP6038 (Olokizumab) 240 mg q4w | RA0083 CDP6038 (Olokizumab) 60 mg q2w | RA0083 CDP6038 (Olokizumab) 60 mg q4w | RA0083 Placebo
Number analyzed (Participants) | 10 | 15 | 11 | 14 | 28 | 24
Percentage of subjects | 100.00 | 71.43 | 80.00 | 69.23 | 78.26 | 65.22

23. Secondary Outcome: Percentage of Subjects With DAS28(CRP) ≤3.2 at Week 24 of Study RA0089
Description: DAS28(CRP) was calculated using the TJC and SJC from 28 joints, the PtGADA-VAS, andCRP according to the formula: DAS28(CRP)=0.56 * (TJC)^1/2 + 0.28 * (SJC)^1/2 + 0.36 * ln(CRP[mg/L]+1) + 0.014 * PtGADA + 0.96 Assessments: • TJC and SJC: assessed on same 2-point scale (0=absent; 1=present). • PtGADA: 100 mm VAS (0=very good, no symptoms; 100=very poor, severe symptoms). • CRP value calculated in mg/L. The 28 joints included shoulders, elbows, wrists; MCP, thumb IP, and PIP joints of hands; and knees. Scores on DAS28(CRP) range from 0 to approximately 10, where scores >5.1 correspond with active disease, scores <3.2 correspond with well controlled disease, and scores <2.6 correspond with remission or similar. Percentage of participants with DAS28(CRP) ≤3.2 were reported.
Time Frame: Week 24 (Study RA0089)
Population: as for outcome 6
Measure: Number; unit: Percentage of subjects
Arm/Group | RA0083 CDP6038 (Olokizumab) 120 mg q2w | RA0083 CDP6038 (Olokizumab) 120 mg q4w | RA0083 CDP6038 (Olokizumab) 240 mg q4w | RA0083 CDP6038 (Olokizumab) 60 mg q2w | RA0083 CDP6038 (Olokizumab) 60 mg q4w | RA0083 Placebo
Number analyzed (Participants) | 10 | 15 | 11 | 14 | 28 | 24
Percentage of subjects | 87.50 | 100.00 | 90.00 | 81.82 | 72.73 | 77.27

24. Secondary Outcome: Percentage of Subjects With DAS28(CRP) ≤3.2 at Week 48 of Study RA0089
Description: as for outcome 23
Time Frame: Week 48 (Study RA0089)
Population: as for outcome 6
Measure: Number; unit: Percentage of subjects
Arm/Group | RA0083 CDP6038 (Olokizumab) 120 mg q2w | RA0083 CDP6038 (Olokizumab) 120 mg q4w | RA0083 CDP6038 (Olokizumab) 240 mg q4w | RA0083 CDP6038 (Olokizumab) 60 mg q2w | RA0083 CDP6038 (Olokizumab) 60 mg q4w | RA0083 Placebo
Number analyzed (Participants) | 10 | 15 | 11 | 14 | 28 | 24
Percentage of subjects | 66.67 | 100.00 | 100.00 | 100.00 | 71.43 | 77.78

25. Secondary Outcome: Percentage of Subjects With DAS28(CRP) ≤3.2 at Week 96 of Study RA0089
Description: DAS28(CRP) was calculated using the TJC and SJC from 28 joints, the PtGADA-VAS, andCRP according to the formula: DAS28(CRP)=0.56 * (TJC)^1/2 + 0.28 * (SJC)^1/2 + 0.36 * ln(CRP[mg/L]+1) + 0.014 * PtGADA + 0.96 Assessments: • TJC and SJC: assessed on same 2-point scale (0=absent; 1=present). • PtGADA: 100 mm VAS (0=very good, no symptoms; 100=very poor, severe symptoms). • CRP value calculated in mg/L. The 28 joints included shoulders, elbows, wrists; MCP, thumb IP, and PIP joints of hands; and knees. Scores on DAS28(CRP) range from 0 to approximately 10, where scores >5.1 correspond with active disease, scores <3.2 correspond with well controlled disease, and scores <2.6 correspond with remission or similar. Since the study was terminated early before Week 96, no data was collected and analyzed at the Week 96 and this Outcome Measure has zero total participants analyzed.
Time Frame: Week 96 (Study RA0089)
Reporting Status: Not Posted

26. Secondary Outcome: Change From Baseline (Week 0 of Study RA0083) in the Clinical Disease Activity Index (CDAI) at Week 48 of Study RA0089
Description: CDAI was calculated using the TJC (28 joints), SJC (28 joints), PtGADA-VAS and PhGADA-VAS, according to the following formula: SJC + TJC + PtGADA + PhGADA Assessments: • TJC and SJC: assessed on the same 2-point scale (0=absent; 1=present). • PtGADA: 10 cm VAS (0=very good, no symptoms; 100=very poor, severe symptoms). • PhGADA: 10 cm VAS (0=very good, asymptomatic and no limitation of normal activities; 100=very poor, very severe symptoms which were intolerable and inability to carry out all normal activities). The 28 joints included the shoulders, elbows, wrists; MCP, thumb IP, and PIP joints of the hands; and the knees. Total score range is from 0-100, with the high scores representing high disease activity. A negative change in CDAI score indicates an improvement in disease activity.
Time Frame: Baseline (Week 0 of Study RA0083) and Week 48 (Study RA0089)
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | RA0083 CDP6038 (Olokizumab) 120 mg q2w | RA0083 CDP6038 (Olokizumab) 120 mg q4w | RA0083 CDP6038 (Olokizumab) 240 mg q4w | RA0083 CDP6038 (Olokizumab) 60 mg q2w | RA0083 CDP6038 (Olokizumab) 60 mg q4w | RA0083 Placebo
Number analyzed (Participants) | 3 | 3 | 6 | 4 | 7 | 9
units on a scale | -72.0000 (86.13362) | -108.0256 (77.85787) | -95.1667 (24.41652) | -75.2870 (46.83603) | -94.7363 (54.63562) | -99.9744 (41.83169)

27. Secondary Outcome: Change From Baseline (Week 0 of Study RA0083) CDAI at Week 96 of Study RA0089
Description: CDAI was calculated using the TJC (28 joints), SJC (28 joints), PtGADA-VAS and PhGADA-VAS, according to the following formula: SJC + TJC + PtGADA + PhGADA Assessments: • TJC and SJC: assessed on the same 2-point scale (0=absent; 1=present). • PtGADA: 10 cm VAS (0=very good, no symptoms; 100=very poor, severe symptoms). • PhGADA: 10 cm VAS (0=very good, asymptomatic and no limitation of normal activities; 100=very poor, very severe symptoms which were intolerable and inability to carry out all normal activities). The 28 joints included the shoulders, elbows, wrists; MCP, thumb IP, and PIP joints of the hands; and the knees. Total score range is from 0-100, with the high scores representing high disease activity. A negative change in CDAI score indicates an improvement in disease activity. Since the study was terminated early before Week 96, no data was collected and analyzed at the Week 96 and this Outcome Measure has zero total participants analyzed.
Time Frame: Baseline (Week 0 of Study RA0083) and Week 96 (Study RA0089)
Reporting Status: Not Posted

28. Secondary Outcome: Change From Baseline (Week 0 of Study RA0083) in the Simplified Disease Activity Index (SDAI) at Week 48 of Study RA0089
Description: SDAI was calculated using the TJC (28 joints), SJC (28 joints), PtGADA-VAS, PhGADA-VAS and CRP (mg/dL]), according to the following formula: SJC + TJC + PtGADA + PhGADA + CRP (mg/dL) Assessments: • TJC and SJC: assessed on the same 2-point scale (0=absent; 1=present). • PtGADA: 10 cm VAS (0=very good, no symptoms; 100=very poor, severe symptoms). • PhGADA: 10 cm VAS (0=very good, asymptomatic and no limitation of normal activities; 100=very poor, very severe symptoms which were intolerable and inability to carry out all normal activities). • CRP range was from 0 to 10 mg/dL. The 28 joints included the shoulders, elbows, wrists; MCP, thumb IP, and PIP joints of the hands; and the knees. The SDAI score ranges from 0 to 86, with higher scores representing worse disease. A negative change in SDAI score indicates an improvement in disease activity.
Time Frame: Baseline (Week 0 of Study RA0083) and Week 48 (Study RA0089)
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | RA0083 CDP6038 (Olokizumab) 120 mg q2w | RA0083 CDP6038 (Olokizumab) 120 mg q4w | RA0083 CDP6038 (Olokizumab) 240 mg q4w | RA0083 CDP6038 (Olokizumab) 60 mg q2w | RA0083 CDP6038 (Olokizumab) 60 mg q4w | RA0083 Placebo
Number analyzed (Participants) | 3 | 3 | 6 | 4 | 7 | 9
units on a scale | -75.6667 (90.23488) | -130.6923 (97.08073) | -125.1667 (48.85659) | -93.7870 (61.23550) | -113.3077 (53.87161) | -127.8633 (38.49694)

29. Secondary Outcome: Change From Baseline (Week 0 of Study RA0083) in the SDAI at Week 96 of Study RA0089
Description: SDAI was calculated using the TJC (28 joints), SJC (28 joints), PtGADA-VAS, PhGADA-VAS and CRP (mg/dL]), as per formula: SJC + TJC + PtGADA + PhGADA + CRP (mg/dL) Assessments: • TJC and SJC: assessed on the same 2-point scale (0=absent; 1=present). • PtGADA: 10 cm VAS (0=very good, no symptoms; 100=very poor, severe symptoms). • PhGADA: 10 cm VAS (0=very good, asymptomatic and no limitation of normal activities; 100=very poor, very severe symptoms which were intolerable and inability to carry out all normal activities). • CRP range was from 0 to 10 mg/dL. The 28 joints included the shoulders, elbows, wrists; MCP, thumb IP, and PIP joints of the hands; and the knees. SDAI score ranges from 0 to 86, with higher scores representing worse disease. A negative change in SDAI score indicates an improvement in disease activity. Since the study was terminated early before Week 96, no data was collected and analyzed at the Week 96 and this Outcome Measure has zero total participants analyzed.
Time Frame: Baseline (Week 0 of Study RA0083) and Week 96 (Study RA0089)
Reporting Status: Not Posted

30. Secondary Outcome: Plasma Concentration of CDP6038 (Olokizumab) at Weeks 4, 8, 12, 16, 24, 32, 40, 48, 72, 96, 120
Description: The CDP6038 (olokizumab) plasma levels data were not collected and analyzed. This Outcome Measure therefore has zero total participants analyzed.
Time Frame: Weeks 4, 8, 12, 16, 24, 32, 40, 48, 72, 96, 120
Reporting Status: Not Posted

31. Secondary Outcome: Plasma Concentration of Anti-CDP6038 (Olokizumab) Antibodies at Weeks 4, 8, 12, 16, 24, 32, 40, 48, 72, 96 and 120
Description: as for outcome 30
Time Frame: Weeks 4, 8, 12, 16, 24, 32, 40, 48, 72, 96, 120
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: From Baseline (Week 0 of Study RA0089) until 30 days after the last dose (maximum up to 562 days)
Description: Reported TEAEs included adverse events that started or worsened after the first dose of CDP6038 (olokizumab) in Study RA0089 and within 30 days after the last dose.
Arm/Group | RA0083 CDP6038 (Olokizumab) 120 mg q2w | RA0083 CDP6038 (Olokizumab) 120 mg q4w | RA0083 CDP6038 (Olokizumab) 240 mg q4w | RA0083 CDP6038 (Olokizumab) 60 mg q2w | RA0083 CDP6038 (Olokizumab) 60 mg q4w | RA0083 Placebo
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/15 | 0/11 | 0/15 | 0/28 | 0/24
Serious Adverse Events (participants affected / at risk) | 1/10 | 0/15 | 2/11 | 2/15 | 5/28 | 4/24
Other Adverse Events (participants affected / at risk) | 8/10 | 13/15 | 10/11 | 12/15 | 25/28 | 21/24
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | RA0083 CDP6038 (Olokizumab) 120 mg q2w (N=10) | RA0083 CDP6038 (Olokizumab) 120 mg q4w (N=15) | RA0083 CDP6038 (Olokizumab) 240 mg q4w (N=11) | RA0083 CDP6038 (Olokizumab) 60 mg q2w (N=15) | RA0083 CDP6038 (Olokizumab) 60 mg q4w (N=28) | RA0083 Placebo (N=24)
Haemorrhoids (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Subdural haematoma (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Duodenal ulcer haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Non-Hodgkin's lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Infectious pleural effusion (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pulmonary tuberculosis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Ligament rupture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Avulsion fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hepatic enzyme increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Epiglottitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Femoral neck fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Third nerve paralysis (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Spondylitic myelopathy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | RA0083 CDP6038 (Olokizumab) 120 mg q2w (N=10) | RA0083 CDP6038 (Olokizumab) 120 mg q4w (N=15) | RA0083 CDP6038 (Olokizumab) 240 mg q4w (N=11) | RA0083 CDP6038 (Olokizumab) 60 mg q2w (N=15) | RA0083 CDP6038 (Olokizumab) 60 mg q4w (N=28) | RA0083 Placebo (N=24)
Coagulopathy (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypocomplementaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
Abnormal sensation in eye (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Asthenopia (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cataract (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Conjunctival haemorrhage (Eye disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Conjunctivitis (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dry eye (Eye disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Vision blurred (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Punctate keratitis (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Aphthous stomatitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (2) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 1 (1)
Dental caries (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 4 (5) | 2 (2)
Enterocolitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Food poisoning (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastritis erosive (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gingival swelling (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haemorrhoids (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Ischaemic enteritis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Mouth ulceration (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 1 (1)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
Stomatitis (Gastrointestinal disorders) | 3 (3) | 2 (2) | 3 (8) | 1 (3) | 2 (3) | 2 (3)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Chest pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Discomfort (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Injection site erythema (General disorders) | 2 (17) | 2 (3) | 1 (4) | 0 (0) | 2 (7) | 2 (3)
Injection site haemorrhage (General disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Injection site induration (General disorders) | 2 (16) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Injection site pruritus (General disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Injection site reaction (General disorders) | 0 (0) | 2 (4) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Injection site swelling (General disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Malaise (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Oedema peripheral (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hepatic function abnormal (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 3 (3)
Hepatic steatosis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 3 (3)
Liver disorder (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypersensitivity (Immune system disorders) | 0 (0) | 0 (0) | 1 (8) | 0 (0) | 0 (0) | 0 (0)
Seasonal allergy (Immune system disorders) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Bronchitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 2 (3) | 0 (0)
Candida infection (Infections and infestations) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
Cystitis (Infections and infestations) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 3 (3) | 1 (1)
Endometritis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Furuncle (Infections and infestations) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 1 (1) | 3 (3) | 2 (2) | 1 (1) | 0 (0)
Gastroenteritis norovirus (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Herpes zoster (Infections and infestations) | 0 (0) | 3 (3) | 1 (1) | 2 (2) | 0 (0) | 1 (1)
Hordeolum (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Influenza (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Localised infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Nasopharyngitis (Infections and infestations) | 3 (6) | 6 (6) | 2 (2) | 6 (7) | 9 (12) | 8 (14)
Onychomycosis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Oral herpes (Infections and infestations) | 1 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Paronychia (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 3 (5) | 0 (0)
Pharyngitis (Infections and infestations) | 0 (0) | 1 (2) | 3 (3) | 1 (2) | 0 (0) | 0 (0)
Pulpitis dental (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tinea pedis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 3 (3)
Tinea versicolour (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 3 (5) | 0 (0) | 1 (1) | 2 (3) | 3 (8)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Arthropod sting (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Bone contusion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chillblains (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 2 (2) | 2 (3) | 1 (1) | 0 (0) | 2 (2) | 1 (1)
Epicondylitis (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Excoriation (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hand fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Laceration (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Ligament sprain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nail avulsion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Thermal burn (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Alanine aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 5 (5)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 5 (6)
Bacterial test positive (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood cholesterol increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Complement factor abnormal (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Low density lipoprotein increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Neutrophil count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
White blood cell count decreased (Investigations) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Diabetes mellitus (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypercholesterolaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
Hyperlipidaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Atlantoaxial instability (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Coccydynia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (2)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Periarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Spinal ligament ossification (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tendonitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
Carpal tunnel syndrome (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 2 (4) | 0 (0) | 0 (0) | 2 (2) | 2 (2) | 4 (11)
Hyperaesthesia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Breast mass (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Menopausal symptoms (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (3) | 1 (1) | 2 (3) | 3 (5) | 1 (1)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 4 (4) | 1 (1)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Upper respiratory tract inflammation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 1 (2)
Alopecia (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 1 (1) | 0 (0)
Dermatitis bullous (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dermatitis psoriasiform (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Eczema (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Eczema asteatotic (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Hyperkeratosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Miliaria (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 2 (2)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (2) | 1 (1) | 1 (1) | 4 (4) | 0 (0)
Seborrhoeic dermatitis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin ulcer (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (2)
Swelling face (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 2 (2) | 2 (2)

LIMITATIONS AND CAVEATS:
The clinical trial was terminated early following a strategic UCB decision to out-license the study drug for further development. No data were collected at Week 96 or beyond; no analysis was performed on study drug plasma levels or antibodies.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. The Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.